CLINICAL TRIAL: NCT00324818
Title: Therapy and Prevention for Sexually Associated Bacterial Vaginosis
Brief Title: Treatment of Bacterial Vaginosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Jane Schwebke, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R01AI048044 (NIH)
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Bacterial Vaginosis
Keywords: bacterial vaginosis; treatment
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Metronidazole; Azithromycin

INTERVENTIONS:
Drug: metronidazole and azithromycin

SUMMARY:
We are trying to determine if longer duration of therapy with metronidazole or combination therapy of metronidazole plus azithromycin results in better cure rates for BV

DETAILED DESCRIPTION:
Bacterial vaginosis (BV) is the most prevalent cause of symptomatic vaginal discharge in the U.S. and has been associated with complications including preterm delivery of infants, pelvic inflammatory disease (PID), urinary tract infections (UTI) and acquisition/transmission of sexually transmitted diseases (STDs) including human immunodeficiency virus (HIV). Control of BV has been advocated for decreasing the prevalence of these complications. The etiology of BV remains unknown and the current treatment regimens are inadequate in terms of initial cure and recurrence rates. Further, half of all women who meet the clinical diagnostic criteria for BV are asymptomatic and treatment of these women remains controversial. More detailed characterization of the origins, natural history and response to therapy would supply data to guide control efforts. We will approach these problems through a multifaceted interdisciplinary evaluation of women with and without BV.

The specific aims {and hypotheses} of this project are:

1. To conduct studies to determine optimal agents and duration of therapy for BV {Hypothesis: Longer duration of therapy and combination therapy will result in higher cure rates and lower recurrence rates of BV; response to therapy differs between women with asymptomatic BV and symptomatic BV}
2. To examine the role of condoms in the prevention of BV {Hypothesis: BV is a sexually transmitted infection, thus recurrence rates of BV will be lower among women with higher condom usage rates}
3. To further explore the role of Mobiluncus spp., organisms strongly associated with the syndrome, by utilizing specimens derived from the above studies.

{Hypothesis: Mobiluncus is involved in the pathogenesis of BV at least in a subset of women, and the persistence of this organism is associated with lack of cure and recurrence of BV}

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic bacterial vaginosis

Exclusion Criteria:

* Pregnancy
* Other genital infections

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600
Dates: Start 2002-07; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
cure of bacterial vaginosis (BV)
  percent of women without BV at follow up

CONTACTS AND LOCATIONS:
Overall Officials: Jane Schwebke, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Jefferson County Department of Health STD Clinic, Birmingham, Alabama, United States